CLINICAL TRIAL: NCT02676284
Title: Study of the Clinical and Biomechanical Effectiveness of Durolane SJ in Rhizarthrosis
Brief Title: Durolane SJ for Treatment of Rhizarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zambon SAU (Industry)
Collaborators: Bioventus LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DURE04
Record Dates: First submitted 2016-01-20; First posted 2016-02-08 (Estimated); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Rhizarthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Durolane SJ (Experimental): single dose injection. One infiltration of the study product in the trapeziometacarpal (TMC) joint. The study treatment contains sodium hyaluronate 20 mg/mL, in a 1 mL prefilled syringe.
  Interventions: Device: Durolane SJ

INTERVENTIONS:
Device: Durolane SJ — DUROLANE® is a clear, transparent, viscous gel of highly purified, stabilized, non-animal-derived sodium hyaluronate that is biosynthesized using bacterial fermentation. NASHA technology is used to stabilize naturally entangled hyaluronic acid (HA) chains to produce a gel. The gel is suspended in phosphate-buffered saline at a concentration of 20 mg/mL .

SUMMARY:
The main objective of the trial is to assess the clinical changes in terms of physical examination, VAS Scale and the Quick-DASH questionnaire, and the biomechanical parameters in terms of mobility of the TMC joint, the grip strength of the hand and lateral pinch strength in patients with rhizarthrosis after administration of viscosupplementation.

The secondary objectives of the trial will be to assess the safety of the treatment with viscosupplementation, and the correlation between the clinical and biomechanical changes at the end of the trial.

DETAILED DESCRIPTION:
This is a prospective, open, non-comparative study in 36 subjects with rhizarthrosis, comparing signs and symptoms before and after a single injection of DUROLANE SJ in the affected hand.

Subjects were assessed pre-treatment and at 1, 3, and 6 months post-treatment. This study is associated with a post marketing commitment with the European Notified Body, BSI, to confirm DUROLANE SJ's effectiveness in rhizarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes aged 18 to 75 years.
* Diagnosis of Grade II-III rhizarthrosis in either hand, according to the criteria of Eaton and Littler.
* TMC joint pain lasting longer than 6 months and baseline pain value greater than or equal to 4 on the VAS scale (0 to 10) and less than 4 in the contralateral hand joint if there is pain.

Exclusion Criteria:

* Anticoagulant medication
* Rheumatic disease involving the wrist, hand and fingers, such as rheumatoid arthritis or gout
* Active rheumatoid arthritis
* Previous surgery of the hand
* Systemic infectious processes
* Neoplastic disease
* Subjects with contraindications to hyaluronic acid
* Subjects with known hypersensitivity to hyaluronic acid or any of the components of the preparation under study
* Previous hyaluronic acid injections in the hand
* Subjects likely to miss the clinical follow-up visits
* Taking of analgesics 24 hours before scheduled clinical assessments
* Pregnant subjects
* Any condition that in the opinion of the physician recommends exclusion of the subject

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eloisa Velasco Ruiz, MD, Principal Investigator — Hospital Sant Joan Despi Moises Broggi
Locations (3):
- Spain (3):
  - Hospital Sant Joan Despi Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Corporació Sanitària Parc Taulí, Barcelona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 patients will take part in the trial. Being a pilot trial, it is considered that the "n" will allow us to adequately assess the clinical and biomechanical changes in order to calculate the suitable "n" for a trial with a larger "n". Patients will be recruited from 3 centres and the recruitment of patients between centres will be competitive
Pre-assignment Details: All subjects were assigned to the same study treatment.
Groups:
- DUROLANE SJ: Sodium hyaluronate, 20 mg/mL, single injection
Period: Overall Study
Arm/Group | DUROLANE SJ
Started | 36
Completed | 35
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety Set = all subjects who received any exposure to study treatment (injection). One patients of the enrolled set discontinued before injection hence was not considered in the safety set.
Arm/Group | DUROLANE SJ
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (61.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 5
Region of Enrollment [Number; unit: participants]
  Spain | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Measured by the VAS Scale
Description: Visual Analogue Scale (VAS) pain in injected hand. The VAS scale ranges from 0 cm (least pain) to 10 cm (most pain).
  A Visual Analogue Scale (VAS) is a measurement instrument that measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
Time Frame: Baseline and 26 weeks
Population: Full Analysis Set: Safety Set subjects with at least 1 post injection visit effectiveness assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | DUROLANE SJ
Number analyzed (Participants) | 35
units on a scale | -2.00 (0.28)

2. Secondary Outcome: Change From Baseline in Biomechanical Function, Measured by the Quick DASH Questionnaire
Description: The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities.This is a self-report questionnaire that patients can use to rate difficulty and interference with daily life. Quick DASH questionnaire is a shortened version of the DASH Outcome Measure which uses 11 items to measure physical function and symptoms in people with musculoskeletal disorders of the upper limb. Possible scores range from 11-55, which can be remapped to a 0-100 scale. This latter ranges from 0 units (most functionality) to 100 units (least functionality).
Time Frame: Baseline and 26 weeks
Population: Full Analysis Set: Safety Set subjects with at least 1 post injection visit effectiveness assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | DUROLANE SJ
Number analyzed (Participants) | 35
units on a scale | -10.8 (2.36)

ADVERSE EVENTS:
Time Frame: Throughout the study, up to 24 weeks.
Arm/Group | DUROLANE SJ
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 4/35
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DUROLANE SJ (N=35)
Pain (General disorders) | 3 (3)
Swelling (General disorders) | 1 (1)
Post Inflammation (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No